CLINICAL TRIAL: NCT01127542
Title: A Single Arm Phase II Study to Investigate the Use of Lenalidomide in the Treatment of Patients With Early Stage CLL Associated With Poor Prognostic Factors
Brief Title: RESPeCT: Revlimid Early Stage Poor Prognosis Chronic Lymphocytic Leukaemia (CLL) Trial
Acronym: RESPeCT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Potential safety issue of second primary malignancies in patients treated with lenalidomide.
Sponsor: The Christie NHS Foundation Trust (Other)
Collaborators: Celgene Corporation (Industry); Leukemia Research Fund (Other)
Responsible Party: Angela Ball, R&D manager, The Christie NHS Foundation Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09_DOG06_99; 2009-011078-14 (EudraCT Number); ISRCTN (Registry Identifier: ISRCTN84606869)
Record Dates: First submitted 2010-05-19; First posted 2010-05-21 (Estimated); Last update posted 2011-12-05 (Estimated); Status verified 2011-12

CONDITIONS: Chronic Lymphocytic Leukaemia
MeSH Terms: conditions — Leukemia, B-Cell | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lenalidomide for early stage poor prognosis CLL (Experimental)
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide — Daily oral lenalidomide. Starting dose of 2.5mg daily, escalating to target dose of 10mg daily.
  Other Names: Revlimid; CC-5013

SUMMARY:
The majority of patients with CLL are diagnosed with early stage disease (Binet stage A or Rai stage 0/I). Standard management of such patients is observation, and with median age at diagnosis of 72 and median time to progression of >5-10 years, many will never require treatment. In contrast, a proportion of patients have more aggressive disease, and over the last decade, a number of molecular factors have been identified that may be used to identify patients with poor prognosis disease . Each is associated with shortened time to treatment (typically less than 3 years in patients with 2 of more factors), reduced survival, with in the case of p53/ATM inactivation, resistance to treatment. Whether it is possible to improve the outcome of patients with CLL and adverse prognostic factors by early intervention with treatment is unknown. Several trials in the 1980's demonstrated that treatment of stage A CLL with conventional chemotherapy (chlorambucil) did not alter the natural history of the disease, although none of these studies stratified patients according to risk. The choice of alternative potential therapeutic agents is limited; they should be effective in patients with adverse prognostic factors, have acceptable toxicity, be able to overcome the drug resistance associated with p53/ATM inactivation and ideally be orally administered. Two recent phase II trials have demonstrated that Lenalidomide is effective in the treatment of relapsed/refractory disease. Importantly, both studies included a high proportion of patients with adverse prognostic factors including p53 inactivation. The principle objective of this study is to investigate the efficacy of Lenalidomide in achieving disease response (complete remission and clearance of minimal residual disease) in patients with poor risk early stage disease, together with assessment of safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Binet stage A CLL
* 2 or more risk factors:
* Unmutated IgVH locus (≥98% homology to germline sequence)
* CD38 expression (>7%)
* Deletion of chromosome 11q22 (>20% by FISH)
* Deletion of chromosome 17p13 (>10% by FISH)
* Over 18 years old
* Capable to provide written informed consent
* ECOG performance status < 2
* Life expectancy > 2 years
* Must agree to not share lenalidomide with someone else
* Must agree not to donate blood whilst taking the study drug and for one week after discontinuation of treatment.
* Female subjects of childbearing potential and all male subjects must agree to comply with the stipulations of the pregnancy prevention plan.

Exclusion Criteria:

* Current or recent (within the last 1 month) participation in another clinical trial investigating the action of an investigational medicinal product for the treatment of CLL
* Pregnant or lactating
* Known positivity for human immunodeficiency virus (HIV) types 1 or 2
* Prior history of malignancies, other than CLL, unless the subject was treated with curative intent and has been free of the disease for ≥3 years. Exceptions include the following:
* Basal cell carcinoma of the skin
* Squamous cell carcinoma of the skin
* Carcinoma in situ of the cervix
* Carcinoma in situ of the breast
* Significantly abnormal renal or hepatic function (creatinine clearance < 60ml/min, serum aspartate aminotransferase (AST) > 3 x upper limit of normal (ULN), serum bilirubin > 34μmol/l)
* Laboratory tumour lysis syndrome according to the Cairo-Bishop classification. Subjects may be enrolled when these abnormalities have been corrected.
* Peripheral neuropathy (grade ≥ 2)
* Previous treatment for CLL
* Previous treatment with Thalidomide or immunomodulatory derivative drugs (including Lenalidomide)
* Treatment with corticosteroids (for CLL or other indications) < 28 days from study entry
* Evidence of Richter's transformation
* Unsupported absolute neutrophil count < 1x109/l or platelet count < 50x10*9/l not due to CLL
* Active autoimmune haemolytic anaemia or thrombocytopenia
* Any other medical or psychological condition that in the view of the investigator would be likely to impact compliance with the protocol or interfere with trial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2010-05; Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Complete Remission with clearance of Minimal Residual Disease (MRD) | 6 months (or earlier if clinically indicated)

SECONDARY OUTCOMES:
Event free survival | Treatment/ progression/ death details collected at all visits (6 visits per month in dose escalation, 1 visit per month in dose maintenance, annual in long-term follow-up)
  Defined as interval from the first treatment day to the first sign of disease progression, treatment for relapse or death (whichever occurs first).
Safety & tolerability of treatment (occurrence of adverse events) | Assessed at all visits (6 visits per month in dose escalation, 1 visit per month in dose maintenance, annual in long-term follow-up)
  Adverse events will be monitored according to NCI CTCAE v3 from screening until 1 month after treatment discontinuation/ trial closure. Adverse event data will be captured at all visits (6 visits per month in dose escalation, 1 visit per month in dose maintenance). Adverse event data will be assessed by blood tests, physical exam/ vital signs and pregnancy testing.
Time to next treatment | Treatment details collected at all visits (6 visits per month in dose escalation, 1 visit per month in dose maintenance, annual in long-term follow-up)
  Defined as interval between first treatment day on the study protocol to the first day of the next course of CLL therapy following disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Bloor, Principal Investigator — The Christie NHS Foundation Trust
Locations (9):
- United Kingdom (9):
  - The Royal Bournemouth Hospital, Bournemouth, Dorset
  - Heart of England NHS Foundation Trust, Birmingham
  - Addenbrooke's Hospital, Cambridge
  - University Hospital of Wales, Cardiff
  - St James's University Hospital, Leeds
  - The Royal Liverpool and Broadgreen University Hospital, Liverpool
  - King's College Hospital, London
  - The Christie NHS Foundation Trust, Manchester
  - Mid Yorkshire Hospitals NHS Trust, Wakefield